CLINICAL TRIAL: NCT02409654
Title: Randomized Controlled Trial of Tailored Stroke Prevention Strategy for Newly Diagnosed Atrial Fibrillation From a Targeted Screening Program Using Handheld Single-lead ECG Device
Brief Title: Hong Kong Outpatient AF Screening Using Single-lead ECG Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HK-OPD-AF
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized stroke prevention (Active Comparator): (i) Patient education (ii) Assess individual risk of stroke using the CHADS2 and CHA2DS2VASc score and risk of major bleeding using the HAS-BLED score (iii) Recommendation of evidence-based stroke prevention therapy based on international guidelines (iv) Patient audit and follow-up (v) Patients not on appropriate OAC without adequate explanation will be referred to Cardiology Outpatient Clinic for second opinion
  Interventions: Other: Patient education; Other: Routine care
- Routine Care (Placebo Comparator): The iECG tracing and report is provided to the attending doctor. Prescription of OAC is left to the discretion of the attending doctor.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Patient education — (i) Patient education (ii) Assess individual risk of stroke using the CHADS2 and CHA2DS2VASc score and risk of major bleeding using the HAS-BLED score (iii) Recommendation of evidence-based stroke prevention therapy based on international guidelines (iv) Patient audit and follow-up (v) Patients not on appropriate OAC without adequate explanation will be referred to Cardiology Outpatient Clinic for second opinion
  Arms: Individualized stroke prevention
Other: Routine care — The iECG tracing and report is provided to the attending doctor. Prescription of OAC is left to the discretion of the attending doctor.

SUMMARY:
Stroke is a leading cause of mortality, morbidity and rising healthcare cost worldwide. In 'real-world' practice, AF is often diagnosed too late at time of stroke and detection can be difficult because AF may be present without symptoms and intermittent in nature. Furthermore, utilization of adequate oral anticoagulation therapy (OAC) for stroke prevention is suboptimal in Hong Kong. The challenge is to identify AF prior to occurrence of stroke. The latest European guidelines recommend opportunistic screening for people >=65 years by pulse palpation followed by 12-lead ECG. However, 12-lead ECG requires a trained technician, time consuming, requires the patient to lie on an examination couch and is not readily available in most outpatient clinics in Hong Kong. A practical screening test is needed. Our study aims to evaluate the feasibility, acceptability and incremental cost of an outpatient based AFscreening program using the AliveCor device. Newly diagnosed AF patients will be randomized to routine care versus individualized stroke prevention strategy which consists of patient education, stroke and bleeding risk assessment, evidence-based OAC recommendation, patient audit and follow-up to improve OAC utilization for stroke prevention. We envisage this study will provide timely evidence to inform policy decisions concerning population-based AF-screening for AF for stroke prevention.

DETAILED DESCRIPTION:
Study Design

The study consists of 2 stages. The screening study examines the feasibility of screening to identify undiagnosed AF in the elderly (>=65 years) using a validated hand-held ECG device and the impact of screening on clinical and economic outcomes at the population level. Subsequent intervention study is a randomized-controlled study comparing an individualized stroke prevention strategy with routine care to prevent stroke in screen-detected AF patients.

Stage 1: AF Screening Study

Screening will be performed in 2 Cardiology and 4 Family Medicine Specialty Out-Patient Clinics (SOPC) at a tertiary referral hospital in Hong Kong. Subjects who meet inclusion and exclusion criteria will sign informed consent for Stage 1 and 2 studies separately, prior to conducting ECG screening.

Stage 2: Randomized Study of Individualized Stroke Prevention vs. Routine Care

Intervention

Screen detected AF patients (new or known AF) from Stage 1 who are not already receiving appropriate OAC for stroke prevention who signed informed consent are randomized 1:1 to routine care or an individualized stroke prevention strategy. Participants will be randomized using block randomization method to assure both groups have the same number of subjects.

Individualized Stroke Prevention Strategy

(i) Patient education on AF and stroke risk. (ii) Assess individual risk of stroke using the CHADS2 and CHA2DS2VASc score and risk of major bleeding using the HAS-BLED score (iii) Recommendation of evidence-based stroke prevention therapy (iv) Patient audit and follow-up: Patients not on appropriate OAC without adequate explanation will be referred to Cardiology SOPC for second opinion.

Routine Care

The iECG tracing and report is provided to the attending doctor. Prescription of OAC is left to the discretion of the attending doctor.

Follow-up

Participants will be followed prospectively every 12 months up to 3 years for clinical events including death, ischemic stroke, any thromboembolic events, intracranial and other major bleeding and stroke prevention therapy. Screen-detected AF patients from Stage 1 who declined to participate in the intervention study will be followed up in a registry.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or over

Exclusion Criteria:

* Severe coexisting medical condition that would prevent participation (eg, dementia, terminal illness)
* Inability to read/understand the consent form and participation information statement

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Utilization rates of evidence-based stroke prevention therapy | 3 years

SECONDARY OUTCOMES:
Rates of newly diagnosed atrial fibrillation in elderly >65 years of age | 3 years
Clinical outcomes including death, stroke and bleeding | 12 months
Patient awareness questionnaire | 12 months
Incremental cost per new AF case detected | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P Yan, MBBS, FACC, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

REFERENCES:
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Background] Mant J, Fitzmaurice DA, Hobbs FD, Jowett S, Murray ET, Holder R, Davies M, Lip GY. Accuracy of diagnosing atrial fibrillation on electrocardiogram by primary care practitioners and interpretative diagnostic software: analysis of data from screening for atrial fibrillation in the elderly (SAFE) trial. BMJ. 2007 Aug 25;335(7616):380. doi: 10.1136/bmj.39227.551713.AE. Epub 2007 Jun 29. PMID 17604299
- [Background] Hobbs FD, Fitzmaurice DA, Mant J, Murray E, Jowett S, Bryan S, Raftery J, Davies M, Lip G. A randomised controlled trial and cost-effectiveness study of systematic screening (targeted and total population screening) versus routine practice for the detection of atrial fibrillation in people aged 65 and over. The SAFE study. Health Technol Assess. 2005 Oct;9(40):iii-iv, ix-x, 1-74. doi: 10.3310/hta9400. PMID 16202350
- [Background] Sudlow M, Rodgers H, Kenny RA, Thomson R. Identification of patients with atrial fibrillation in general practice. BMJ. 1999 Jan 23;318(7178):264. doi: 10.1136/bmj.318.7178.264. No abstract available. PMID 9915750
- [Background] Bjorck S, Palaszewski B, Friberg L, Bergfeldt L. Atrial fibrillation, stroke risk, and warfarin therapy revisited: a population-based study. Stroke. 2013 Nov;44(11):3103-8. doi: 10.1161/STROKEAHA.113.002329. Epub 2013 Aug 27. PMID 23982711
- [Background] Lee VW, Tam CS, Yan BP, Man Yu C, Yin Lam Y. Barriers to warfarin use for stroke prevention in patients with atrial fibrillation in Hong Kong. Clin Cardiol. 2013 Mar;36(3):166-71. doi: 10.1002/clc.22077. Epub 2012 Nov 14. PMID 23151816
- [Background] Koponen L, Rekola L, Ruotsalainen T, Lehto M, Leino-Kilpi H, Voipio-Pulkki LM. Patient knowledge of atrial fibrillation: 3-month follow-up after an emergency room visit. J Adv Nurs. 2008 Jan;61(1):51-61. doi: 10.1111/j.1365-2648.2007.04465.x. PMID 18173735
- [Background] Smith MB, Christensen N, Wang S, Strohecker J, Day JD, Weiss JP, Crandall BG, Osborn JS, Anderson JL, Horne BD, Muhlestein JB, Lappe DL, Moss H, Oliver J, Viau K, Bunch TJ. Warfarin knowledge in patients with atrial fibrillation: implications for safety, efficacy, and education strategies. Cardiology. 2010;116(1):61-9. doi: 10.1159/000314936. Epub 2010 May 26. PMID 20502012
- [Background] Court H, Greenland K, Margrain TH. Measuring patient anxiety in primary care: Rasch analysis of the 6-item Spielberger State Anxiety Scale. Value Health. 2010 Sep-Oct;13(6):813-9. doi: 10.1111/j.1524-4733.2010.00758.x. Epub 2010 Jun 17. PMID 20561315
- [Background] Marjoram J, Strachan R, Allan A, Allan E. Screening for colorectal cancer: a general-practice-based study. Br J Gen Pract. 1996 May;46(406):283-86. PMID 8762743